CLINICAL TRIAL: NCT04170725
Title: Muscular and Cutaneous Dysfunction in Postural Tachycardia Syndrome
Brief Title: Muscular and Cutaneous Dysfunction in POTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POTS
Record Dates: First submitted 2019-11-12; First posted 2019-11-20 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Postural Tachycardia Syndrome
Keywords: POTS
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients and Healthy volunteers (Experimental): Patients and Healthy volunteers will undergo a 14-day training protocol. No study drugs will be administered. Patients and Healthy volunteers will be instructed regarding their training protocol. Training sessions will be undertaken on days 1, 3, 5, 7, 9 and 11 after the first examination day. Participants will be asked to contract their TA muscle repeatedly by pulling the right foot towards the head in a standing position while the heel remains on the ground (at 5 second intervals). In order to carry out the training they will also receive a video demonstrating the exercise. On days 1 and 3 they will do the exercise for 5 minutes, on days 5 and 7 for 10 minutes and on days 9 and 11 for 15 minutes.
  Interventions: Other: Patient and Healthy Volunteers training protocol

INTERVENTIONS:
Other: Patient and Healthy Volunteers training protocol — Patients and Healthy Volunteers will undergo a 14-day endurance training protocol. No study drugs will be administered. Patients and Healthy Volunteers will be instructed regarding their training protocol. Training sessions will be undertaken on days 1, 3, 5, 7, 9 and 11 after the first examination day. Patients and Healthy Volunteers will be asked to contract their TA muscle repeatedly by pulling the right foot towards the head in a standing position while the heel remains on the ground (at 5 second intervals). In order to carry out the training they will also receive a video demonstrating the exercise. On days 1 and 3 they will do the exercise for 5 minutes, on days 5 and 7 for 10 minutes and on days 9 and 11 for 15 minutes.

SUMMARY:
POTS patients seem to experience orthostasis-dependent muscle weakness and pain as well as increased muscle fatigue upon physical activity, which can be improved by regular aerobic exercise. However, reduced sweat production of the extremities with limited control of the body temperature leads to exercise intolerance, so that sticking to a training program becomes a challenge for most patients. Recordings of MVRCs provide a new tool to assess muscle membrane dysfunction, depending on ischemia, surface temperature and training. As muscle dysfunction is assumed to be present in the majority of POTS patients but has not yet been scientifically studied the present study aims at understanding the muscular and cutaneous functioning in POTS using MVRC recordings, dependent both on orthostatic stress and exercise training as well as body temperature regulation. Our main hypothesis is that POTS patients experience functional muscle dysfunction that may be linked to altered muscle perfusion or body temperature regulation.

The purpose of this study is to examine muscular and cutaneous dysfunction in POTS in order to i) better understand the underlying pathology for symptoms and to ii) ultimately improve treatment options.

DETAILED DESCRIPTION:
POTS patients seem to experience orthostasis-dependent muscle weakness and pain as well as increased muscle fatigue upon physical activity, which can be improved by regular aerobic exercise. However, reduced sweat production of the extremities with limited control of the body temperature leads to exercise intolerance, so that sticking to a training program becomes a challenge for most patients. Recordings of MVRCs provide a new tool to assess muscle membrane dysfunction, depending on ischemia, surface temperature and training. As muscle dysfunction is assumed to be present in the majority of POTS patients but has not yet been scientifically studied the present study aims at understanding the muscular and cutaneous functioning in POTS using MVRC recordings, dependent both on orthostatic stress and exercise training as well as body temperature regulation. Our main hypothesis is that POTS patients experience functional muscle dysfunction that may be linked to altered muscle perfusion or body temperature regulation.

The purpose of this study is to examine muscular and cutaneous dysfunction in POTS in order to i) better understand the underlying pathology for symptoms and to ii) ultimately improve treatment options.

The study includes two examination days with the same procedure for all participants. In between the examination days, participants will undergo an endurance training protocol for 14 days. The first examination day takes place in two parts: Participants will first receive repetitive MVRC recordings of the right tibialis anterior muscle (TA): 1) before, during and after repetitive stimulation of the right TA (intermittent 20Hz for 10 min) in the supine position. Then MVRC recordings will be done from the left TA 2) in the supine position and during the 60° HUT upright position for 10 minutes. The duration of this first part is approximately 60 minutes. The second part consists of a TST of the hands and feet only, including a SWT on the index, middle and ring finger of both hands. This second part also lasts about 60 minutes. On the second examination day, the first part (only 1)) of the first examination day will be repeated. In between the examination days training sessions will be undertaken on days 1, 3, 5, 7, 9 and 11 between the examination days. Participants will be asked to contract their TA muscle repeatedly by pulling the right foot towards the head in a standing position while the heel remains on the ground (at 5 second intervals). In order to carry out the training they will also receive a video demonstrating the exercise. On days 1 and 3 they will do the exercise for 5 minutes, on days 5 and 7 for 10 minutes and on days 9 and 11 for 15 minutes.

ELIGIBILITY:
Inclusion Criteria Patients:

* Informed consent as documented by signature
* Patients with diagnosed neuropathic POTS
* Age: ≥18 years and ≤ 60 years

Inclusion Criteria Healthy Volunteers:

* Informed consent as documented by signature
* Age: ≥18 years and ≤ 60 years

Exclusion Criteria Patients:

* Pregnancy and breastfeeding
* Inability to adhere to the training protocol

Exclusion Criteria Healthy Volunteers:

* Pregnancy and breastfeeding
* Intake of vasoactive medication or known, non-treated arterial hypertension
* Inability to adhere to the training protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Change of early supernormality in% | Day 14
  Change of early super normality as the most important parameter of MVRC measurements during HUT and fatigue in patients with neuropathic POTS compared to healthy subjects.

SECONDARY OUTCOMES:
Change of relative refractory period in msec | Day 14
  During HUT and muscle fatigue
Change of late supernormality period in % | Day 14
  During HUT and muscle fatigue
Change of early supernormality % after Muscle endurance training | Day 14
  Muscle endurance training induced changes of MVRC measurements
Change of relative refractory period in msec after Muscle endurance training | Day 14
  Muscle endurance training induced changes of MVRC measurements
Change of late supernormality in % after Muscle endurance training | Day 14
  Muscle endurance training induced changes of MVRC measurements
Area of palmar sweat production (in cm2) | Day 1
  Qualitative sweat production
Area of plantar sweat production (in cm2) | Day 1
  Qualitative sweat production
Skin wrinkling grade | Day 1
  Skin wrinkling grade
Intramuscular and skin temperature change | Day 14
  Intramuscular and skin temperature changes during HUT and fatigue
Recapillarization time at the lower extremities | Day 14
  Recapillarization time at the lower extremities before and during HUT
Heart rate changes | Day 14
  Heart rate changes during HUT and fatigue
Blood pressure changes | Day 14
  Blood pressure changes during HUT and fatigue
Maximal Tibialis Anterior peak force and endurance time | Day 14
  Maximal Tibialis Anterior peak force and endurance time before and after training
Circumference of the lower legs | Day 14
  Circumference of the lower legs before and after training

CONTACTS AND LOCATIONS:
Overall Officials: Werner Z'Graggen, MD, Principal Investigator — Inselspital Bern, Department of Neurosurgery & Neurology
Locations (1):
- Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson JW, Lambert EA, Sari CI, Dawood T, Esler MD, Vaddadi G, Lambert GW. Cognitive function, health-related quality of life, and symptoms of depression and anxiety sensitivity are impaired in patients with the postural orthostatic tachycardia syndrome (POTS). Front Physiol. 2014 Jun 25;5:230. doi: 10.3389/fphys.2014.00230. eCollection 2014. PMID 25009504
- [Background] Boerio D, Z'Graggen WJ, Tan SV, Guetg A, Ackermann K, Bostock H. Muscle velocity recovery cycles: effects of repetitive stimulation on two muscles. Muscle Nerve. 2012 Jul;46(1):102-11. doi: 10.1002/mus.23267. PMID 22692998
- [Background] Bostock H, Baumann C, Humm AM, Z'graggen WJ. Temperature dependency of human muscle velocity recovery cycles. Muscle Nerve. 2012 Aug;46(2):264-6. doi: 10.1002/mus.23429. PMID 22806376
- [Background] Bostock H, Campero M, Serra J, Ochoa J. Velocity recovery cycles of C fibres innervating human skin. J Physiol. 2003 Dec 1;553(Pt 2):649-63. doi: 10.1113/jphysiol.2003.046342. Epub 2003 Sep 8. PMID 12963801
- [Background] Deb A, Morgenshtern K, Culbertson CJ, Wang LB, Hohler AD. A survey-based analysis of symptoms in patients with postural orthostatic tachycardia syndrome. Proc (Bayl Univ Med Cent). 2015 Apr;28(2):157-9. doi: 10.1080/08998280.2015.11929217. PMID 25829642
- [Background] Freeman R, Wieling W, Axelrod FB, Benditt DG, Benarroch E, Biaggioni I, Cheshire WP, Chelimsky T, Cortelli P, Gibbons CH, Goldstein DS, Hainsworth R, Hilz MJ, Jacob G, Kaufmann H, Jordan J, Lipsitz LA, Levine BD, Low PA, Mathias C, Raj SR, Robertson D, Sandroni P, Schatz I, Schondorff R, Stewart JM, van Dijk JG. Consensus statement on the definition of orthostatic hypotension, neurally mediated syncope and the postural tachycardia syndrome. Clin Auton Res. 2011 Apr;21(2):69-72. doi: 10.1007/s10286-011-0119-5. No abstract available. PMID 21431947
- [Background] Freeman R, Wieling W, Axelrod FB, Benditt DG, Benarroch E, Biaggioni I, Cheshire WP, Chelimsky T, Cortelli P, Gibbons CH, Goldstein DS, Hainsworth R, Hilz MJ, Jacob G, Kaufmann H, Jordan J, Lipsitz LA, Levine BD, Low PA, Mathias C, Raj SR, Robertson D, Sandroni P, Schatz IJ, Schondorf R, Stewart JM, van Dijk JG. Consensus statement on the definition of orthostatic hypotension, neurally mediated syncope and the postural tachycardia syndrome. Auton Neurosci. 2011 Apr 26;161(1-2):46-8. doi: 10.1016/j.autneu.2011.02.004. Epub 2011 Mar 9. No abstract available. PMID 21393070
- [Background] Fu Q, Levine BD. Exercise in the postural orthostatic tachycardia syndrome. Auton Neurosci. 2015 Mar;188:86-9. doi: 10.1016/j.autneu.2014.11.008. Epub 2014 Nov 21. PMID 25487551
- [Background] Fu Q, Levine BD. Exercise and non-pharmacological treatment of POTS. Auton Neurosci. 2018 Dec;215:20-27. doi: 10.1016/j.autneu.2018.07.001. Epub 2018 Jul 4. PMID 30001836
- [Background] Grubb BP. Postural tachycardia syndrome. Circulation. 2008 May 27;117(21):2814-7. doi: 10.1161/CIRCULATIONAHA.107.761643. No abstract available. PMID 18506020
- [Background] Humm AM, Bostock H, Troller R, Z'Graggen WJ. Muscle ischaemia in patients with orthostatic hypotension assessed by velocity recovery cycles. J Neurol Neurosurg Psychiatry. 2011 Dec;82(12):1394-8. doi: 10.1136/jnnp-2011-300444. Epub 2011 Jun 7. PMID 21653205
- [Background] Jacob G, Costa F, Shannon JR, Robertson RM, Wathen M, Stein M, Biaggioni I, Ertl A, Black B, Robertson D. The neuropathic postural tachycardia syndrome. N Engl J Med. 2000 Oct 5;343(14):1008-14. doi: 10.1056/NEJM200010053431404. PMID 11018167
- [Background] Jacob G, Diedrich L, Sato K, Brychta RJ, Raj SR, Robertson D, Biaggioni I, Diedrich A. Vagal and Sympathetic Function in Neuropathic Postural Tachycardia Syndrome. Hypertension. 2019 May;73(5):1087-1096. doi: 10.1161/HYPERTENSIONAHA.118.11803. PMID 30879357
- [Background] Lambert E, Lambert GW. Sympathetic dysfunction in vasovagal syncope and the postural orthostatic tachycardia syndrome. Front Physiol. 2014 Jul 28;5:280. doi: 10.3389/fphys.2014.00280. eCollection 2014. PMID 25120493
- [Background] Masuki S, Eisenach JH, Schrage WG, Johnson CP, Dietz NM, Wilkins BW, Sandroni P, Low PA, Joyner MJ. Reduced stroke volume during exercise in postural tachycardia syndrome. J Appl Physiol (1985). 2007 Oct;103(4):1128-35. doi: 10.1152/japplphysiol.00175.2007. Epub 2007 Jul 12. PMID 17626834
- [Background] Schondorf R, Low PA. Idiopathic postural orthostatic tachycardia syndrome: an attenuated form of acute pandysautonomia? Neurology. 1993 Jan;43(1):132-7. doi: 10.1212/wnl.43.1_part_1.132. PMID 8423877
- [Background] Sheldon RS, Grubb BP 2nd, Olshansky B, Shen WK, Calkins H, Brignole M, Raj SR, Krahn AD, Morillo CA, Stewart JM, Sutton R, Sandroni P, Friday KJ, Hachul DT, Cohen MI, Lau DH, Mayuga KA, Moak JP, Sandhu RK, Kanjwal K. 2015 heart rhythm society expert consensus statement on the diagnosis and treatment of postural tachycardia syndrome, inappropriate sinus tachycardia, and vasovagal syncope. Heart Rhythm. 2015 Jun;12(6):e41-63. doi: 10.1016/j.hrthm.2015.03.029. Epub 2015 May 14. No abstract available. PMID 25980576
- [Background] Shibata S, Fu Q, Bivens TB, Hastings JL, Wang W, Levine BD. Short-term exercise training improves the cardiovascular response to exercise in the postural orthostatic tachycardia syndrome. J Physiol. 2012 Aug 1;590(15):3495-505. doi: 10.1113/jphysiol.2012.233858. Epub 2012 May 28. PMID 22641777
- [Background] Tan SV, Z'graggen WJ, Boerio D, Rayan DL, Howard R, Hanna MG, Bostock H. Membrane dysfunction in Andersen-Tawil syndrome assessed by velocity recovery cycles. Muscle Nerve. 2012 Aug;46(2):193-203. doi: 10.1002/mus.23293. PMID 22806368
- [Background] Tan SV, Z'Graggen WJ, Boerio D, Rayan DR, Norwood F, Ruddy D, Howard R, Hanna MG, Bostock H. Chloride channels in myotonia congenita assessed by velocity recovery cycles. Muscle Nerve. 2014 Jun;49(6):845-57. doi: 10.1002/mus.24069. Epub 2014 May 2. PMID 24037712
- [Background] Wilder-Smith EP, Guo Y, Chow A. Stimulated skin wrinkling for predicting intraepidermal nerve fibre density. Clin Neurophysiol. 2009 May;120(5):953-8. doi: 10.1016/j.clinph.2009.03.011. Epub 2009 Apr 16. PMID 19375384
- [Background] Z'Graggen WJ, Aregger F, Farese S, Humm AM, Baumann C, Uehlinger DE, Bostock H. Velocity recovery cycles of human muscle action potentials in chronic renal failure. Clin Neurophysiol. 2010 Jun;121(6):874-81. doi: 10.1016/j.clinph.2010.01.024. Epub 2010 Feb 23. PMID 20181515
- [Background] Z'graggen WJ, Bostock H. Velocity recovery cycles of human muscle action potentials and their sensitivity to ischemia. Muscle Nerve. 2009 May;39(5):616-26. doi: 10.1002/mus.21192. PMID 19229874
- [Background] Z'Graggen WJ, Brander L, Tuchscherer D, Scheidegger O, Takala J, Bostock H. Muscle membrane dysfunction in critical illness myopathy assessed by velocity recovery cycles. Clin Neurophysiol. 2011 Apr;122(4):834-41. doi: 10.1016/j.clinph.2010.09.024. Epub 2010 Nov 1. PMID 21044861
- [Background] Z'Graggen WJ, Trautmann JP, Bostock H. Force training induces changes in human muscle membrane properties. Muscle Nerve. 2016 Jun;54(1):144-6. doi: 10.1002/mus.25149. PMID 27104654
- [Background] Z'graggen WJ, Troller R, Ackermann KA, Humm AM, Bostock H. Velocity recovery cycles of human muscle action potentials: repeatability and variability. Clin Neurophysiol. 2011 Nov;122(11):2294-9. doi: 10.1016/j.clinph.2011.04.010. Epub 2011 May 8. PMID 21555240
- [Background] Ziemssen T, Siepmann T. The Investigation of the Cardiovascular and Sudomotor Autonomic Nervous System-A Review. Front Neurol. 2019 Feb 12;10:53. doi: 10.3389/fneur.2019.00053. eCollection 2019. PMID 30809183